CLINICAL TRIAL: NCT00263887
Title: Multi-center, Randomized Trial With I.V. Prolastin® to Evaluate Frequency of Exacerbations and Progression of Emphysema by Means of Multi-slice CT Scans in Patients With Congenital Alpha-1-antitrypsin Deficiency.
Brief Title: Alpha-1-Antitrypsin (AAT) To Treat Emphysema In AAT-Deficient Patients (EXACTLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100533
Record Dates: First submitted 2005-09-12; First posted 2005-12-09 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha 1 proteinase inhibitor; alpha1 proteinase inhibitor; congenital emphysema; replacement therapy
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Congenital lobar emphysema | interventions — alpha 1-Antitrypsin; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Prolastin
  Interventions: Drug: Alpha1-Proteinase Inhibitor (Human)
- Group 2 (Placebo Comparator)
  Interventions: Drug: Albumin (Human) 20%, United States Pharmacopeia (USP)

INTERVENTIONS:
Drug: Alpha1-Proteinase Inhibitor (Human) — Weekly infusion of 60 mg/kg body weight for 2 years
  Other Names: Prolastin; alpha-1 antitrypsin (AAT); BAY x 5747; BAY 10-5233; TAL-05-00007; NDC 13533-601-30; NDC 13533-601-35
  Arms: Group 1
Drug: Albumin (Human) 20%, United States Pharmacopeia (USP) — Weekly infusion for 2 years. Albumin (Human) 20% will be diluted with 5% glucose to a final concentration of 2.0%.
  Other Names: Plasbumin®-20; Plasbumin®-20 (Low Aluminum); Albumin (Human) 20%; TAL-05-00008; TAL-05-00024; BAY 34-9255; NDC 3533-683-20; NDC 1533-683-71; NDC 13533-691-20; NDC 13533-691-71
  Arms: Group 2

SUMMARY:
The goal of this trial was to explore the utility of evaluating emphysema progression through CT scans measuring lung density during a 2 year period of weekly infusions of either placebo or human alpha-1-antitrypsin (AAT; Prolastin®). Exacerbation data recorded in patient diaries were also collected. All efficacy data were analyzed for potential use in evaluating Prolastin efficacy in this and other clinical trials.

DETAILED DESCRIPTION:
This is a one to one randomized, placebo-controlled, clinical, exploratory study with the aim of collecting information on possible clinical endpoints i.e., the progression of emphysema by lung density measurements with CT scan and frequency of exacerbations that could be used for a subsequent placebo controlled clinical trial. Progression of disease will be investigated in 80 patients with alpha-1-antitrypsin deficiency, who will be treated with human alpha-1-antitrypsin (AAT; Prolastin®) or placebo weekly for two years to analyze the effect of treatment on lung density and exacerbations. Targeted augmentation therapy with weekly infusions of Prolastin® will be a dose of 60 mg/kg body weight (range of 51.72 to 71.43 mg per kg body weight).

Therefore, this study focuses on several questions:

* Is the 15th percentile point calculated by analysis of CT lung histograms a useful endpoint for clinical trials in AAT deficiency?
* Is quantitation of exacerbations in AAT-deficient patients a useful endpoint for clinical trials in AAT deficiency?
* Are there significant differences between the treatments in favor of Prolastin®?

ELIGIBILITY:
Inclusion Criteria:

* Patient with pulmonary emphysema due to severe congenital AAT deficiency of phenotype protease inhibitor Z (PiZ) or other rare genotypes (not MS, MZ or SZ) and AAT serum level < 11 microns (µM) or < 80 mg/dL (status to be confirmed by phenotyping and genotyping)
* Inspiratory capacity (VC - ERV) > 1.2 L and forced expiratory volume at one second (FEV1) < 80% of predicted value post bronchodilator
* FEV1/VC < 70% of predicted value post-bronchodilator or transfer factor of carbon monoxide (KCO) < 80% of predicted value post-bronchodilator
* History of at least one exacerbation in the past 2 years
* Written informed consent

Exclusion Criteria:

* FEV1 < 25% of predicted value post-bronchodilator
* Augmentation therapy for more than one month with plasma-derived human alpha 1-antitrypsin (AAT) within the last 2 years
* History of lung transplant
* Any lung surgery within the past 2 years
* On any thoracic surgery waiting list
* Diagnosis of liver cirrhosis
* Severe concomitant disease
* Active pulmonary infection/exacerbations within the last month
* Active smoking during the last 6 months or plasma positive for cotinine
* Body weight < 42 kg or > 92 kg
* Pregnancy or lactation
* Women of child-bearing potential without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asger Dirksen, MD PHD, Principal Investigator — University of Copenhagen
Locations (3):
- Gentofte Hospital Department of Respiratory Medicine, Hellerup, Denmark
- Department of Pulmonary Medicine, Malmö University Hospital, Malmo, Sweden
- Queen Elizabeth Hospital, Birmingham, England, United Kingdom

REFERENCES:
- [Result] Brand P, Schulte M, Wencker M, Herpich CH, Klein G, Hanna K, Meyer T. Lung deposition of inhaled alpha1-proteinase inhibitor in cystic fibrosis and alpha1-antitrypsin deficiency. Eur Respir J. 2009 Aug;34(2):354-60. doi: 10.1183/09031936.00118408. Epub 2009 Feb 27. PMID 19251783
- [Result] Dirksen A, Piitulainen E, Parr DG, Deng C, Wencker M, Shaker SB, Stockley RA. Exploring the role of CT densitometry: a randomised study of augmentation therapy in alpha1-antitrypsin deficiency. Eur Respir J. 2009 Jun;33(6):1345-53. doi: 10.1183/09031936.00159408. Epub 2009 Feb 5. PMID 19196813
- [Result] Soriano JB, Miravitlles M. Your racing horses will help you to quit: a lesson for COPD and alpha1-antitrypsin deficiency research. Eur Respir J. 2009 Jun;33(6):1244-6. doi: 10.1183/09031936.00026409. No abstract available. PMID 19483042
- [Derived] Vijayasaratha K, Stockley RA. Relationship between frequency, length, and treatment outcome of exacerbations to baseline lung function and lung density in alpha-1 antitrypsin-deficient COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:789-96. doi: 10.2147/COPD.S31797. Epub 2012 Nov 27. PMID 23226015
- [Derived] Carter RI, Mumford RA, Treonze KM, Finke PE, Davies P, Si Q, Humes JL, Dirksen A, Piitulainen E, Ahmad A, Stockley RA. The fibrinogen cleavage product Aalpha-Val360, a specific marker of neutrophil elastase activity in vivo. Thorax. 2011 Aug;66(8):686-91. doi: 10.1136/thx.2010.154690. Epub 2011 May 26. PMID 21617168
- [Derived] Stockley RA, Parr DG, Piitulainen E, Stolk J, Stoel BC, Dirksen A. Therapeutic efficacy of alpha-1 antitrypsin augmentation therapy on the loss of lung tissue: an integrated analysis of 2 randomised clinical trials using computed tomography densitometry. Respir Res. 2010 Oct 5;11(1):136. doi: 10.1186/1465-9921-11-136. PMID 20920370
- [Derived] Parr DG, Dirksen A, Piitulainen E, Deng C, Wencker M, Stockley RA. Exploring the optimum approach to the use of CT densitometry in a randomised placebo-controlled study of augmentation therapy in alpha 1-antitrypsin deficiency. Respir Res. 2009 Aug 13;10(1):75. doi: 10.1186/1465-9921-10-75. PMID 19678952
- See also: FDA Approved Product Labeling Information - Prolastin® — http://www.talecris-pi.info/inserts/Prolastin.pdf
- See also: FDA Approved Product Labeling Information - Plasbumin®-20 (Low Aluminum) — http://www.talecris-pi.info/inserts/plasbumin20la.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study with 3 sites in Denmark, Sweden, and the United Kingdom.
Period: Overall Study
Arm/Group | Prolastin (60 mg/kg Body Weight) | Placebo
Started | 38 | 39
Completed | 35 | 32
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lung transplantation | 1 | 2
Not completed — Too ill to attend visit | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Disease progression | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolastin (60 mg/kg Body Weight) | Placebo | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 34 | 67
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.68 (8.29) | 55.26 (9.68) | 54.97 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 36
  Male | 25 | 16 | 41
Region of Enrollment [Number; unit: participants]
  Denmark | 18 | 17 | 35
  United Kingdom | 12 | 14 | 26
  Sweden | 8 | 8 | 16
Severity of COPD at baseline [Number; unit: participants] — Severity of Chronic Obstructive pulmonary Disease (COPD) at baseline according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) classes
  participants
    None | 2 | 2 | 4
    Mild | 1 | 2 | 3
    Moderate | 10 | 8 | 18
    Severe | 19 | 20 | 39
    Very Severe | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Progression Rate of Emphysema Determined by Change in 15th Percentile of Lung Density Measured by Annual CT Scan of the Whole Lung
Time Frame: 24 or 30 months
Population: The modified Intent-To-Treat Population was defined as all subjects in the Intent-To-Treat (ITT) Population (all randomized subjects) who had a valid baseline CT scan and at least one valid post-baseline CT scan measurement.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Prolastin (60 mg/kg Body Weight) | Placebo
Number analyzed (Participants) | 35 | 32
g/L
  Baseline | 47.980 (19.072) | 45.477 (16.949)
  Endpoint | 45.085 (19.433) | 41.354 (16.260)
  Change from Baseline | -2.895 (4.739) | -4.124 (4.147)
Statistical Analysis 1: Comparison: Prolastin (60 mg/kg Body Weight) vs Placebo; The main effect ANCOVA model includes the change from baseline to endpoint as the dependent variable, treatment and center as fixed factors, change in logarithm of total lung volume and baseline measurement as covariates; Test type: Superiority or Other; p = 0.049, ANCOVA

2. Secondary Outcome: Change in Lung Density at Each Visit as Measured by Computed Tomography
Time Frame: 24 or 30 months
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: g/L

3. Secondary Outcome: The Frequency of Exacerbations as Determined by Patient Diary.
Time Frame: 24 or 30 months
Reporting Status: Not Posted

4. Secondary Outcome: The Deterioration of the Lung Function Will be Assessed by Measurement of the Change in Forced Expiratory Volume at One Second (FEV1) and Transfer Factor of Carbon Monoxide (KCO)
Time Frame: 24 or 30 months
Reporting Status: Not Posted

5. Secondary Outcome: Duration and Severity of the Exacerbations
Time Frame: 24 or 30 months
Reporting Status: Not Posted

6. Secondary Outcome: Mortality
Time Frame: 24 or 30 months
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life With a Disease Specific Instrument, the St. George's Respiratory Questionnaire
Time Frame: 24 or 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Prolastin (60 mg/kg Body Weight) | Placebo
Serious Adverse Events (participants affected / at risk) | 9/38 | 15/39
Other Adverse Events (participants affected / at risk) | 37/38 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prolastin (60 mg/kg Body Weight) (N=38) | Placebo (N=39)
Atrial fibrillation (Cardiac disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4
Malaria (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epixtaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prolastin (60 mg/kg Body Weight) (N=38) | Placebo (N=39)
Angina pectoris (Cardiac disorders) | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Gastritis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Pyrexia (General disorders) | 3 | 2
Chest pain (General disorders) | 2 | 5
Infusion related reaction (General disorders) | 2 | 0
Oedema (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 5
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 4
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Seasonal allergy (Immune system disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 24 | 22
Pneumonia (Infections and infestations) | 12 | 9
Sinusitis (Infections and infestations) | 5 | 5
Influenza (Infections and infestations) | 4 | 3
Tooth abscess (Infections and infestations) | 3 | 5
Bronchitis (Infections and infestations) | 2 | 1
Localised infection (Infections and infestations) | 2 | 1
Oral candidiasis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 3
Eye infection (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 5
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 2
Blood potassium decreased (Investigations) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Monoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Headache (Nervous system disorders) | 9 | 10
Dizziness (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 1 | 2
Sinus headache (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 2 | 2
Phlebitis (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed within thirty days and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution, which satisfies both parties.